CLINICAL TRIAL: NCT06310005
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Subcutaneous Doses and Multiple Subcutaneous Doses Over 6 Weeks of BI 3006337 in Healthy Male Japanese Subjects (Single-blind, Randomised Within Dose Groups, Placebo-controlled, Parallel Group Design)
Brief Title: A Study in Healthy Japanese Men to Test How Well Different Doses of BI 3006337 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1466-0003
Record Dates: First submitted 2024-03-08; First posted 2024-03-13 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Trial consists of a single-rising dose (SRD) and multiple dose (MD) part. In SRD part, the groups will be dosed consecutively in ascending order. The decision proceeding to MD part will be based upon safety and tolerability of all the preceding dose groups in SRD part. Within each dose group, patients will be randomized to either BI 3006337 or placebo.
Who Masked: Participant
Masking Description: The trial is designed single-blind. The treatments administered (BI 3006337 or placebo) will be blinded to subjects but will be known to the investigators (outcome assessors).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (SRD) (Placebo Comparator): Participants received one single dose of Placebo matching BI 3006337, as subcutaneous injection on Day 1 of the single-rising dose part.
  Interventions: Drug: Placebo
- Single-rising dose part (SRD): BI 3006337 low dose (Experimental): Participants received one single low dose of BI 3006337 as subcutaneous injection on Day 1 of the single-rising dose part.
  Interventions: Drug: BI 3006337
- SRD part: BI 3006337 medium dose (Experimental): Participants received one single medium dose of BI 3006337 as subcutaneous injection on Day 1 of the single-rising dose part.
  Interventions: Drug: BI 3006337
- SRD part: BI 3006337 high dose (Experimental): Participants received one single high dose of BI 3006337 as subcutaneous injection on Day 1 of the single-rising dose part.
  Interventions: Drug: BI 3006337
- Placebo (MD) (Placebo Comparator): Participants received one dose of Placebo matching BI 3006337, as subcutaneous injection once per week for 6 weeks (multiple dose part (MD)).
  Interventions: Drug: Placebo
- Multiple dose part (MD): BI 3006337 high dose (Experimental): Participants received one high dose of BI 3006337 as subcutaneous injection once per week for 6 weeks (multiple dose part (MD)).
  Interventions: Drug: BI 3006337

INTERVENTIONS:
Drug: BI 3006337 — BI 3006337
  Arms: Multiple dose part (MD): BI 3006337 high dose; SRD part: BI 3006337 high dose; SRD part: BI 3006337 medium dose; Single-rising dose part (SRD): BI 3006337 low dose
Drug: Placebo — Placebo
  Arms: Placebo (MD); Placebo (SRD)

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of BI 3006337 in healthy male subjects following s.c. administration of single rising doses and multiple doses over 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Japanese ethnicity, according to the following criteria: born in Japan, have lived outside of Japan < 10 years, and have parents and grandparents who are Japanese
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 25.0 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Conference of Harmonization - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Subjects who agree to minimise the risk of making their partner pregnant by fulfilling any of the following criteria starting from the start of injection of trial medication until 30 days after end of injection of trial medication:

  * Use of adequate contraception, any of the following methods plus condom: intrauterine device, combined oral contraceptives that started at least 2 months prior to the first drug administration
  * Vasectomized (vasectomy at least 1 year prior to enrolment)
  * Surgical sterilization (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner
  * Female partner is postmenopausal, defined as no menses for 1 year without an alternative medical cause

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimeter of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or PR outside the range of 50 to 90 bpm at screening visit
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Hospital Tokyo, Tokyo, Shinjuku-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The purpose of this study was to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single rising subcutaneous doses and multiple subcutaneous doses over 6 weeks of BI 3006337 in healthy male Japanese subjects (single-blind, randomised within dose groups, placebo controlled, parallel group design).
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all patients as required.
Groups:
- Single-rising Dose Part (SRD): BI 3006337 50 mg Dose: Participants received one single 50 milligrams (mg) dose of BI 3006337 as subcutaneous injection on Day 1 of the single-rising dose part.
- SRD Part: BI 3006337 100 mg Dose: Participants received one single 100 mg dose of BI 3006337 as subcutaneous injection on Day 1 of the single-rising dose part.
- SRD Part: BI 3006337 150 mg Dose: Participants received one single 150 mg dose of BI 3006337 as subcutaneous injection on Day 1 of the single-rising dose part.
- Multiple Dose Part (MD): BI 3006337 150 mg Dose: Participants received one 150 mg dose of BI 3006337 as subcutaneous injection once per week for 6 weeks (multiple dose part (MD)).
Period: Overall Study
Arm/Group | Placebo (SRD) | Single-rising Dose Part (SRD): BI 3006337 50 mg Dose | SRD Part: BI 3006337 100 mg Dose | SRD Part: BI 3006337 150 mg Dose | Placebo (MD) | Multiple Dose Part (MD): BI 3006337 150 mg Dose
Started | 6 | 6 | 6 | 6 | 3 | 9
Completed | 6 | 6 | 6 | 6 | 3 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all participants who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (SRD) | Single-rising Dose Part (SRD): BI 3006337 50 mg Dose | SRD Part: BI 3006337 100 mg Dose | SRD Part: BI 3006337 150 mg Dose | Placebo (MD) | Multiple Dose Part (MD): BI 3006337 150 mg Dose | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (6.7) | 34.5 (10.9) | 28.2 (9.1) | 27.7 (8.1) | 31.3 (10.1) | 31.4 (8.8) | 30.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 3 | 9 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 3 | 9 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 6 | 3 | 9 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: Number of participants with treatment-emergent adverse events (TEAE) is presented.
Time Frame: SRD part: From BI 3006337 administration until end of residual effect period (REP), 3 weeks. MD part: From first until last BI 3006337 administration + REP, up to 9 weeks.
Population: Treated set (TS): The treated set included all participants who were treated with at least one dose of trial drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (SRD) | Single-rising Dose Part (SRD): BI 3006337 50 mg Dose | SRD Part: BI 3006337 100 mg Dose | SRD Part: BI 3006337 150 mg Dose | Placebo (MD) | Multiple Dose Part (MD): BI 3006337 150 mg Dose
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9
Participants | 4 | 4 | 2 | 2 | 0 | 8

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 3006337 in Serum Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of BI 3006337 in serum over the time interval from 0 extrapolated to infinity (AUC0-inf) is presented.
Time Frame: Within 3 hours (hrs) before BI 3006337 administration and at 1.5, 3, 7, 11, 15, 23, 27, 31, 35, 39, 47, 58, 72, 96, 120, 168, 240, 336, 504, and 672 hrs, and at end of trial examination, up to Day 40 after BI 3006337 administration.
Population: Pharmacokinetic parameter analysis set (PKS): This set included all participants in the TS who provided at least one pharmacokinetic (PK) endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliters (h*ng/ml)
Arm/Group | Single-rising Dose Part (SRD): BI 3006337 50 mg Dose | SRD Part: BI 3006337 100 mg Dose | SRD Part: BI 3006337 150 mg Dose
Number analyzed (Participants) | 6 | 6 | 6
hours*nanograms/milliliters (h*ng/ml) | 41400 (35.7) | 61400 (23.1) | 109000 (34.6)

3. Secondary Outcome: Maximum Measured Concentration of BI 3006337 in Serum (Cmax)
Description: Maximum measured concentration of BI 3006337 in serum (Cmax) is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliters (ng/ml)
Arm/Group | Single-rising Dose Part (SRD): BI 3006337 50 mg Dose | SRD Part: BI 3006337 100 mg Dose | SRD Part: BI 3006337 150 mg Dose
Number analyzed (Participants) | 6 | 6 | 6
nanograms/milliliters (ng/ml) | 665 (43.7) | 1050 (78.9) | 1730 (46.4)

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 3006337 in Serum Over the Dosing Interval Tau at Steady State (AUCtau, ss) After the Last Dose in Week 6
Description: Area under the concentration-time curve of BI 3006337 in serum over the dosing interval tau at steady state (AUCtau, ss) after the last dose in Week 6 is presented.
Time Frame: Within 3 hours (hrs) before last BI 3006337 administration and at 3, 7, 11, 15, 23, 27, 31, 35, 39, 47, 72, and 168 hrs after last BI 3006337 administration.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliters (h*ng/ml)
Arm/Group | Multiple Dose Part (MD): BI 3006337 150 mg Dose
Number analyzed (Participants) | 9
hours*nanograms/milliliters (h*ng/ml) | 91600 (41.5)

5. Secondary Outcome: Maximum Measured Concentration of BI 3006337 in Serum at Steady State (Cmax, ss) After the Last Dose in Week 6
Description: Maximum measured concentration of BI 3006337 in serum at steady state (Cmax, ss) after the last dose in Week 6 is presented.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliters (ng/ml)
Arm/Group | Multiple Dose Part (MD): BI 3006337 150 mg Dose
Number analyzed (Participants) | 9
nanograms/milliliters (ng/ml) | 1720 (76.0)

ADVERSE EVENTS:
Time Frame: For on-treatment AEs: From BI 3006337 administration until end of residual effect period (REP), 3 weeks (SRD part). From first until last BI 3006337 administration + REP, up to 9 weeks (MD part). For all-cause mortality: From first drug administration until end of trial (EoT), up to 40 days (SRD) and up to 74 days (MD).
Description: Treated set (TS): The treated set included all participants who were treated with at least one dose of trial drug.
Arm/Group | Placebo (SRD) | Single-rising Dose Part (SRD): BI 3006337 50 mg Dose | SRD Part: BI 3006337 100 mg Dose | SRD Part: BI 3006337 150 mg Dose | Placebo (MD) | Multiple Dose Part (MD): BI 3006337 150 mg Dose
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 2/6 | 2/6 | 0/3 | 8/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (SRD) (N=6) | Single-rising Dose Part (SRD): BI 3006337 50 mg Dose (N=6) | SRD Part: BI 3006337 100 mg Dose (N=6) | SRD Part: BI 3006337 150 mg Dose (N=6) | Placebo (MD) (N=3) | Multiple Dose Part (MD): BI 3006337 150 mg Dose (N=9)
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 5
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Urinary occult blood positive (Investigations) | 0 | 2 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT06310005/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT06310005/SAP_001.pdf